CLINICAL TRIAL: NCT00095212
Title: Androgen Effects in HIV-infected Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Steven Grinspoon, M.D., Principal Investigator, MGH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK54167 (completed); R01DK054167 (NIH)
Record Dates: First submitted 2004-11-01; First posted 2004-11-02 (Estimated); Results first posted 2010-03-15 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infection
Keywords: HIV; women; androgen; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Transdermal Testosterone (Patch) (Active Comparator): 300 micrograms applied twice a week
  Interventions: Drug: 1 Transdermal Testosterone (Patch)
- 2 Placebo Patch (identical in appearance) (Placebo Comparator): placebo patch (0 micrograms of testosterone)applied twice a week
  Interventions: Drug: 2 Placebo Patch

INTERVENTIONS:
Drug: 1 Transdermal Testosterone (Patch) — 300 micrograms twice a week
  Arms: 1 Transdermal Testosterone (Patch)
Drug: 2 Placebo Patch — Placebo patch (0 micrograms of testosterone) applied twice a week
  Arms: 2 Placebo Patch (identical in appearance)

SUMMARY:
Androgen deficiency in HIV-infected women is associated with sarcopenia and may cause critical reductions in physical functioning and reduced bone density. The effects of long-term androgen therapy on lean body mass, bone density and other clinical endpoints including quality of life, functional status and neurocognitive function in HIV-infected women are not known.

DETAILED DESCRIPTION:
We will perform an 18-month randomized, double-blinded, placebo-controlled study among relatively androgen deficient women with HIV, to determine the effects of testosterone administration on lean body mass. The administered dose will be 300 micrograms twice a week vs. identical placebo in the form of a transdermal preparation. Secondary endpoints include effects on bone density, quality of life, neurocognitive function and menstrual function. Open label administration at 300 micrograms twice a week will be initiated for 12 months in all subjects following the randomized portion of the study. Assuming a 15% dropout rate and 25 randomized patients, the probability is 80 percent that the study will detect a treatment difference at a two sided 5.000 percent significance level, if the true difference between the treatments is 2.7 kg. This is based on the assumption that the standard deviation of the response variable, lean body mass by DEXA, is 2.3 kg, as was shown by Choi et al1 over 12 weeks in HIV-infected women at the same dose of 300 ug 2x/week.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 - 55
* BMI less than or equal to 26
* HIV-infected
* Androgen deficient, with free testosterone < 3 pg/mL
* Stable antiretroviral regimen for 3 months prior to study
* Tubal ligation, hysterectomy, or verbalized understanding of appropriate barrier contraception methods. Subjects will be counseled in appropriate barrier contraception methods and the counseling will be documented.

Exclusion Criteria:

* Use of anabolic agent, including testosterone, GH or other preparations within 3 months of the study.
* Use of megestrol acetate within 3 months of the study
* Use of estrogen or any preparation known to affect bone density or bone turnover.This includes oral contraceptives, depo provera or combined progesterone-estrogen injections, and transdermal contraceptive patches.
* Pregnant or breast-feeding
* Hgb < 9.0 mg/dL
* Current participation in another research study conducted by this investigator or past participation in the DHEA study funded by the same grant as this protocol.
* Creatinine > 1.5 mg/dL

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2004-09; Primary Completion 2008-04 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Dolan Looby SE, Collins M, Lee H, Grinspoon S. Effects of long-term testosterone administration in HIV-infected women: a randomized, placebo-controlled trial. AIDS. 2009 May 15;23(8):951-9. doi: 10.1097/QAD.0b013e3283299145. PMID 19287303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in August, 2004 and continued through October, 2006. Subjects were recruited via poster advertisement at community health centers, hospitals, and AIDS Service Organizations, as well as newspaper advertisement and provider referral.
Pre-assignment Details: Prior to randomization at the baseline visit, each subject's doctor was contacted to confirm safety of study enrollment. Subjects age 40 and older were required to have a mammogram performed within one year of study enrollment and provide results. Eligible subjects completed a pregnancy test at each visit and were excluded for a positive test.
Groups:
- Transdermal Testosterone (Patch): 300 micrograms applied twice a week
- Placebo Patch (Identical in Appearance): placebo patch (0 micrograms of testosterone)applied twice a week
Period: Overall Study
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Started | 13 | 12
Completed | 12 | 9
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance) | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45 (2) | 43 (1) | 44 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Lean Body Mass
Description: Represents change in measure from baseline to 18 months. 18 month mean and standard error of the mean for lean body mass measured by dual energy absorptiometry (DEXA)scan.
Time Frame: Baseline (time 0) to 18 months
Population: Responses at 9 and 18 months were pooled as the post treatment repeated measures. All data were included in the analysis, including 9 month data from the 4 subjects who discontinued after the 9 month visit.
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 13 | 12
kilograms | 1.8 (0.5) | 0.8 (0.9)
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); Test type: Superiority or Other; p = 0.04, longitudinal linear mixed effects model

2. Secondary Outcome: Bone Mineral Density of the Hip
Description: Represents change in measure from baseline to 18 months. 18 month mean and standard error of the mean for bone mineral density of the hip measured by dual energy absorptiometry (DEXA)scan.
Time Frame: Baseline (time 0) to 18 months
Measure: Mean (Standard Error); unit: grams per centimeter squared
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 13 | 12
grams per centimeter squared | 0.01 (0.01) | -0.01 (0.01)
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); The study was powered at 80% to detect a significant treatment difference of 2.7 kg in lean body mass between the two groups with 25 randomized patients and a 15% assumed dropout rate, using a two sided 5.0 percent significance level; Test type: Superiority or Other; p = 0.02, Longitudinal linear mixed effects model

3. Secondary Outcome: Quality of Life/Depression: Becks Depression Inventory
Description: Represents change in the mean score from baseline to 18 months. Depression was evaluated with the Beck's Depression Inventory (BDI). The BDI is a 21-item self-report instrument used to assess the presence and severity of symptoms of depression. A Total score in the range of 0-13 is considered minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: Baseline (time 0) to 18 months
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 13 | 12
Units on a scale | -6.8 (2.2) | -1.9 (3.1)
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.02, Longitudinal mixed methods model

4. Secondary Outcome: Quality of Life/Sexual Function: Brief Index of Sexual Function (BISF-W) Domain 7: Problems Affecting Sexual Function
Description: Represents change in measure from baseline to 18 months. The BISF is 22 items with seven domains: Thoughts and Desires, Arousal, Frequency of Sexual Activity, Receptivity/Initiation, Pleasure, Relationship Satisfaction, and Problems Affecting Sexual Function. Data from Domain 7: Problems Affecting Sexual Function is reported. The score range for this domain is -16 to 75,a higher score indicates greater sexual function.
Time Frame: Baseline (time 0) to 18 months
Population: data not available for all subjects as some did not wish to complete the questionnaire
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 9 | 7
Units on a scale | -1.8 (0.8) | 0.5 (0.5)
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.01, Longitudinal mixed methods model

5. Secondary Outcome: Safety: Number of Subjects Reporting a Skin Reaction to the Patch
Description: Represents number of subjects who reported this symptom from baseline to 18 months. Every 6 weeks,subjects were counseled on appropriate barrier contraception methods and a urine pregnancy was performed. Subjects who experienced increased hair growth (facial hair) could remain in the study on a lower dose of testosterone (1 patch per week), but dose reductions were not necessary and full dosing was continued throughout the study for all subjects. Changes in menstrual status, missed periods and/or irregular bleeding, were noted and reported back to the primary care physician if significant.
Time Frame: Baseline (time 0) to 18 months
Measure: Number; unit: participants
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 13 | 12
participants | 4 | 1
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); Test type: Superiority or Other; p = 0.16, Chi-squared

6. Secondary Outcome: Safety: Number of Subjects Reporting a Change in Hair Pattern (Increased Hair on Chin, Upper Lip, Chest, Abdomen, Fore Arms, and Legs)
Description: as for outcome 5
Time Frame: Baseline (time 0) to 18 months
Measure: Number; unit: participants
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 13 | 12
participants | 2 | 4
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); Test type: Superiority or Other; p = 0.29, Chi-squared

7. Secondary Outcome: Safety: Number of Subjects Reporting Acne
Description: as for outcome 5
Time Frame: Baseline (time 0) to 18 months
Measure: Number; unit: participants
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 13 | 12
participants | 4 | 3
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); Test type: Superiority or Other; p = 0.75, Chi-squared

8. Secondary Outcome: Safety: Number of Subjects Reporting a Change in Menstrual Status (Reported More Than One Period in 1 Month or Missed a Period During a Monthly Cycle)
Description: as for outcome 5
Time Frame: Baseline (time 0) to 18 months
Measure: Number; unit: participants
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 13 | 12
participants | 6 | 9
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); Test type: Superiority or Other; p = 0.14, Chi-squared

9. Secondary Outcome: Neurocognitive Function: Hopkins Verbal Learning Test-revised,"Total Recall" Z Score Represents Change in Z Score From Baseline to 18 Months.
Description: This test assesses verbal learning and memory. Subjects are given a list of 12 words and asked to repeat as many words as they can recall during 3 separate trials. The Total Recall Z score is calculated based on the sum of total correct responses for Trials 1,2,& 3. A Z score of 0 equals the 50 percentile, a Z score of 1 is 1 standard deviation above the mean and a Z score of -1 is 1 standard deviation below the mean. The lowest and highest T scores for the HVLT-R are ≤20 and ≥80. This correlates to lowest and highest Z scores of ≤ -3.0 and ≥3.0. A lower Z score is indicative of poor recall.
Time Frame: Baseline (time 0) to 18 months
Population: data not available for all subjects as some did not wish to complete the testing
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 12 | 7
Units on a scale | -0.21 (0.41) | 0.50 (0.37)
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); Test type: Superiority or Other; p = 0.26, t-test, 2 sided

10. Secondary Outcome: Strength: Total Knee Flexion Performed Via Quantitative Muscle Function Testing.
Description: Represents change in isometric force (measured in kilograms) from baseline to 18 months. Peak isometric force of total knee flexion and extension were measured on the best of 2 repetitions for which subjects held a maximum contraction for 5 seconds.
Time Frame: Baseline (time 0) to 18 months
Population: data not available for all subjects due to malfunctioning equipment at some sessions, and some subjects did not wish to complete testing.
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 11 | 8
kilograms | 28.5 (11.0) | 11.0 (4.9)
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); Test type: Superiority or Other; p = 0.22, t-test, 2 sided

11. Secondary Outcome: Strength: Total Knee Extension Performed Via Quantitative Muscle Function Testing.
Description: as for outcome 10
Time Frame: Baseline (time 0) to 18 months
Population: as for outcome 10
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Number analyzed (Participants) | 11 | 9
kilograms | 28.0 (7.6) | 26.9 (10.7)
Statistical Analysis 1: Comparison: Transdermal Testosterone (Patch) vs Placebo Patch (Identical in Appearance); Test type: Superiority or Other; p = 0.94, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected over an 18 month period
Description: Subjects were seen every 6 weeks at which time a physical exam was performed, and subjects reported adverse events and/or safety concerns to the investigator.
Arm/Group | Transdermal Testosterone (Patch) | Placebo Patch (Identical in Appearance)
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/12
Other Adverse Events (participants affected / at risk) | 9/13 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Testosterone (Patch) (N=13) | Placebo Patch (Identical in Appearance) (N=12)
Appendectomy (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject was admitted to the hospital with abdominal pain and underwent surgery. This event is not related to study drug or participation. This subject was receiving testosterone.
ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Subject was seen in the emergency room for discomfort and was diagnosed with an ovarian cyst and uterine fibroid. This event is not related to study participation. Subject was receiving placebo.
uterine fibroid (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Subject was seen in the emergency room for discomfort and was diagnosed with an ovarian cyst and uterine fibroid. This event is not related to study participation. Subject was receiving placebo.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Testosterone (Patch) (N=13) | Placebo Patch (Identical in Appearance) (N=12)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
peripheral neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
candidiasis of the vagina (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sinusitis (Infections and infestations) | 1 (1) | 0 (0)
herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
vertigo (Nervous system disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
simple renal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
excision of bunion (Surgical and medical procedures) | 0 (0) | 1 (1)
elective mammoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No